CLINICAL TRIAL: NCT00852657
Title: Comparison of Surgical Treatment by Tendon Repair and Physiotherapy in the Treatment of Small and Medium-sized Tears of the Rotator Cuff
Brief Title: Comparison of Tendon Repair and Physiotherapy in the Treatment of Small and Medium-sized Tears of the Rotator Cuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Stefan Moosmayer, MD, PhD, Vestre Viken Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 430-04149 (REK)
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff tear; surgical repair; Physiotherapy; Treatment benefit; Surgery
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical treatment (Active Comparator): Open or mini-open tendon repair with acromioplasty
  Interventions: Procedure: Tendon repair with acromioplasty
- Physiotherapy (Active Comparator): Physiotherapy by exercises
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Tendon repair with acromioplasty — Open or mini-open tendon repair in combination with an acromioplasty and eventually a tenodesis of the long head of the biceps
  Arms: Surgical treatment
Procedure: Physiotherapy — According to a rehabilitation program which was established prior to study start.
  Arms: Physiotherapy

SUMMARY:
The purpose of this study is to compare treatment benefits from surgical treatment by tendon repair and from physiotherapy for small and medium-sized rotator cuff tears.

DETAILED DESCRIPTION:
Surgical treatment by tendon repair or physiotherapy are accepted treatment options for small and medium-sized rotator cuff tears, but have never been compared in randomised, controlled studies.

In this study, patients presenting clinical signs together with imaging findings (MRI and sonography) for a full-thickness rotator cuff tear will be randomly allocated to surgery (tendon repair) or physiotherapy. Outcome measuring will be performed by the Constant score, the self report section of the American Shoulder and Elbow Surgeons score (ASES), the Short Form 36 Health Survey (SF-36) and subscores for shoulder motion, pain, strength and patient satisfaction. Scores will be taken at baseline and after 6 months,1, 2, 5, 10 and 15 years by a blinded assessor. All operated shoulders will be controlled by MRI after one year. Patients with no effect from physiotherapy after at least 15 treatment sessions will be offered secondary surgical treatment, and scoring results from last follow-up before surgery will be carried forward to analysis, according to an intention to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history and imaging findings of a rotator cuff tear

Exclusion Criteria:

* Presence of other local or systemic diseases influencing on shoulder function
* History of earlier rotator cuff surgery
* Medical contraindications for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2004-09; Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Constant score | baseline, 6 months, 1, 2, 5, 10, 15 years

SECONDARY OUTCOMES:
self report section of the American Shoulder and Elbow Surgeons score (ASES) | baseline, 6 months, 1, 2, 5, 10, 15 years
Short Form 36 Health Survey (SF-36) | baseline, 6 months, 1, 2, 5, 10, 15 years
Patient satisfaction | 1, 2, 5, 10, 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Moosmayer, MD, Principal Investigator — Vestre Viken Hospital Trust; Hans-Joergen Smith, MD, PhD, Study Chair — University of Oslo, Rikshospitalet
Locations (1):
- Martina Hansen's Hospital, Sandvika, Norway

REFERENCES:
- [Result] Moosmayer S, Lund G, Seljom U, Svege I, Hennig T, Tariq R, Smith HJ. Comparison between surgery and physiotherapy in the treatment of small and medium-sized tears of the rotator cuff: A randomised controlled study of 103 patients with one-year follow-up. J Bone Joint Surg Br. 2010 Jan;92(1):83-91. doi: 10.1302/0301-620X.92B1.22609. PMID 20044684
- [Result] Moosmayer S, Lund G, Seljom US, Haldorsen B, Svege IC, Hennig T, Pripp AH, Smith HJ. Tendon repair compared with physiotherapy in the treatment of rotator cuff tears: a randomized controlled study in 103 cases with a five-year follow-up. J Bone Joint Surg Am. 2014 Sep 17;96(18):1504-14. doi: 10.2106/JBJS.M.01393. PMID 25232074
- [Result] Moosmayer S, Lund G, Seljom US, Haldorsen B, Svege IC, Hennig T, Pripp AH, Smith HJ. At a 10-Year Follow-up, Tendon Repair Is Superior to Physiotherapy in the Treatment of Small and Medium-Sized Rotator Cuff Tears. J Bone Joint Surg Am. 2019 Jun 19;101(12):1050-1060. doi: 10.2106/JBJS.18.01373. PMID 31220021